CLINICAL TRIAL: NCT00848692
Title: B-cell Depletion Using the Monoclonal Anti-CD20 Antibody Rituximab in Chronic Fatigue Syndrome. A Double-blind, Placebo-controlled Study.
Brief Title: Drug Intervention in Chronic Fatigue Syndrome
Acronym: KTS-1-2008
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18257; EudraCT: 2007-007973-22
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2011-06

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic Fatigue Syndrome; CFS; Myalgic Encephalomyelitis; Rituximab; B-lymphocyte depletion; B-cell depletion
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Rituximab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rituximab
  Interventions: Drug: Rituximab
- 2 (Placebo Comparator): Placebo (saline)
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Rituximab — Two infusions of Rituximab 500 mg/m2 (max 1000 mg) given two weeks apart
  Arms: 1
Drug: Saline (NaCl 0,9 %) (placebo) — Two infusions of saline (NaCl 0,9 %) given two weeks apart
  Arms: 2

SUMMARY:
Based on pilot patient observations,the investigators anticipate that chronic fatigue syndrome (CFS) patients may benefit from B-cell depletion therapy.

The hypothesis is that at least a subset of CFS patients have an activated immune system involving B-lymphocytes, and that B-cell depletion may alleviate symptoms.

ELIGIBILITY:
Inclusion Criteria:

* verified chronic fatigue syndrome (CDC-criteria)
* age >18 and <60 years
* informed consent

Exclusion Criteria:

* pregnancy or lactation
* previous malignant disease except basal cell carcinoma of skin and cervical carcinoma in situ
* previous long-term use of immunosuppressive drugs
* previous exposure to rituximab
* endogenous depression
* multi-allergy with risk of serious drug reaction
* reduced renal function (creatinin > 1.2 x UNL)
* reduced liver function (bilirubin or transaminases > 1.5 x UNL)
* known HIV infection
* signs of active viral infection by pretreatment investigations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Symptom alleviation, as compared to baseline, measured by standardized self-reports and quality of life schemes. | 3 months after intervention

SECONDARY OUTCOMES:
Symptom alleviation, as compared to baseline, measured by standardized self-reports and quality of life schemes | 2, 4, 6, 8, 10, 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Olav Mella, MD, PhD, Principal Investigator — Department of Oncology and Medical Physics, Haukeland University Hospital
Locations (1):
- Department of Oncology and Medical Physics, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Fluge O, Bruland O, Risa K, Storstein A, Kristoffersen EK, Sapkota D, Naess H, Dahl O, Nyland H, Mella O. Benefit from B-lymphocyte depletion using the anti-CD20 antibody rituximab in chronic fatigue syndrome. A double-blind and placebo-controlled study. PLoS One. 2011;6(10):e26358. doi: 10.1371/journal.pone.0026358. Epub 2011 Oct 19. PMID 22039471